CLINICAL TRIAL: NCT07299747
Title: A Phase I/IIa Clinical Study Evaluating the Bispecific Antibody-Drug Conjugate VBC103 Targeting Nectin-4 and TROP2 in Subjects With Advanced Malignant Solid Tumors
Brief Title: Clinical Trial of VBC103 in Patients With Advanced Malignant Solid Tumors
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: VelaVigo Bio Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VBC103-01-01
Record Dates: First submitted 2025-12-09; First posted 2025-12-23 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Participants With Advanced Solid Tumor Malignancies

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Phase 1 (Dose Escalation and Backfill)，Phase 2（Dose optimization and Cohort Expansion） (Experimental)
  Interventions: Drug: VBC103

INTERVENTIONS:
Drug: VBC103 — VBC103

SUMMARY:
This study is a multicenter, open-label, multi-dose, first-in-human (FIH) Phase I/IIa study to determine the safety and tolerability of VBC103, as well as the maximum tolerated dose (MTD) and/or recommended Phase II dose (RP2D), PK and further evaluate its efficacy.

ELIGIBILITY:
Inclusion Criteria:

* 1.The subject or their legal representative is willing and able to sign a written ICF before initiating any study procedures.
* 2.Histologically or cytologically confirmed unresectable advanced/metastatic solid tumor that has recurred or progressed during or after standard systemic therapy, or is intolerant to standard therapy, or lacks standard treatment options (applicable only to Phase I and Phase IIa Cohort 5).
* 3.At least one measurable lesion as assessed by the investigator per RECIST v1.1.
* 4.Adult male or female (defined as ≥18 years of age)
* 5.ECOG performance status score of 0-1.
* 6.LVEF ≥50% as measured by ECHO or MUGA within 28 days prior to enrollment.
* 7.Life expectancy exceeding 12 weeks.
* 8.Availability of archived tumor tissue samples or willingness to undergo biopsy sampling.

Exclusion Criteria:

* 1.Any unresolved ≥Grade 2 toxicity from prior anticancer therapy.
* 2.Known active keratitis or corneal ulcer.
* 3.History of interstitial lung disease (e.g., non-infectious interstitial pneumonia, pneumonitis,pulmonary fibrosis, or severe radiation pneumonitis), current interstitial lung disease, or suspected interstitial lung disease based on imaging during the screening period.
* 4.History of underlying pulmonary diseases, including but not limited to pulmonary embolism within 3 months prior to the start of investigational product, severe asthma, severe chronic obstructive pulmonary disease, restrictive lung disease, and other clinically significant pulmonary impairment or requiring supplemental oxygen, as well as any autoimmune, connective tissue, or inflammatory disease involving the lungs (such as rheumatoid arthritis, Sjögren's syndrome, sarcoidosis, etc.) and/or prior pneumonectomy (complete resection).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 255 (Estimated)
Dates: Start 2025-12-04 (Actual); Primary Completion 2027-12-01 (Estimated); Study Completion 2028-12-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of dose-limiting toxicities (DLT) as defined in the protocol | (DLT)From time of first dose of VBC103 to end of DLT period (approximately 21 days)
  Number of patients with at least 1 dose-limiting toxicity (DLT), which is any toxicity defined as a DLT in the Clinical Study Protocol
Incidence of Serious Adverse Events | From time of Informed Consent to 30 days post last dose of VBC103
  Number of patients with serious adverse events by system organ class and preferred term

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | From date of first dose of VBC103 up until progression, or the last evaluable assessment in the absence of progression (approximately 2 years)
  The percentage or number of patients with a confirmed investigator assessed complete or partial response according to response criteria in solid tumours (RECIST v1.1)
Duration of Response (DOR) | From date of first dose of VBC103 up until progression, or the last evaluable assessment in the absence of progression (approximately 2 years)
  The time from date of first response until date of disease progression or last evaluable assessment (RECIST v1.1) in the absence of progression
Disease Control Rate (DCR) at 12 weeks | From date of first dose of VBC103 up until progression, or the last evaluable assessment in the absence of progression (for each patient this is expected to be measured at 12 weeks)
  The percentage of patients with confirmed CR or PR or having SD maintained (RECIST v1.1) for >=11 weeks from first dose
Pharmacokinetics of VBC103: Plasma PK concentrations | From date of first dose of VBC103 up until 30 days post last dose
  Measurement of plasma concentrations of VBC103, total antibody and total unconjugated warhead
Pharmacokinetics of VBC103: Maximum plasma concentration of the study drug (C-max) | From date of first dose of VBC103 up until 30 days post last dose
  Measurement of PK parameters: Maximum observed plasma concentration of the study drug (C-max)
Pharmacokinetics of VBC103: Time to maximum plasma concentration of the study drug (T-max) | From date of first dose of VBC103 up until 30 days post last dose
  Measurement of PK parameters: Time to maximum observed plasma concentration of the study drug (T-max)
Immunogenicity of VBC103: Anti-Drug Antibodies (ADA) | From date of first dose of VBC103 up until 30 days post last dose
  Evaluating the number and percentage of patients who develop Anti-drug antibody (ADA) during treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided